CLINICAL TRIAL: NCT06257134
Title: Impact on Quality of Life of Symptoms Routine E-monitoring Among Dialysis Patients, With Results Notification to Teams. A Cluster Randomised Controlled Trial Nested in a National Registry F-SWIFT (French Symptom Monitoring WIth Feedback Trial)
Brief Title: Impact on Quality of Life of Symptoms Routine E-monitoring Among Dialysis Patients.
Acronym: F-SWIFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Agence de La Biomédecine (Other Government); University of Bordeaux (Other); University Hospital, Bordeaux (Other); University of Sydney (Other); Centre Hospitalier Régional Universitaire de Tours (Other Government); Association France REIN (Unknown); Association AFIDTN (French Association of Dialysis, Transplant and Nephrology Nurses) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023PI052
Record Dates: First submitted 2023-12-23; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: End Stage Renal Disease
Keywords: Symptoms; Quality of life; IPOS-Renal; Dialysis units; ePROMS; Tablets; RedCAP
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: F-SWIFT is a large-scale, multi-center, randomized controlled trial (qualitative and quantitative) nested in a national registry.
  Experimental group
  * Quarterly measurement for 18 months of patients' symptoms using the IPOS-Renal questionnaire, which will be systematically reported to professionals.
  * Measurement every 6 months for 18 months of patients' health-related HRQoL using the EQ-5D-5L, KDQoL-36 and SONG-Fatigue questionnaires.
  Control group
  * No systematic symptom monitoring will be organized, and patients will receive usual care.
  * Measurement of health-related HRQoL every 6 months for 18 months, using the EQ-5D-5L, KDQoL-36 and SONG-Fatigue questionnaires.
  The F-SWIFT project includes a process analysis to underpin the transferability of F-SWIFT in the event of proven effectiveness with a view to large-scale deployment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Patients in the control group will complete three HRQoL questionnaires every six months via a digital tablet during their dialysis session.
  Interventions: Other: No systematic monitoring of symptoms
- Experimental group (Experimental): Every three months, patients in the experimental group will have their symptoms systematically recorded using the IPOS-Renal questionnaire via a digital tablet during their dialysis session.
  Interventions: Other: Systematic monitoring of symptoms

INTERVENTIONS:
Other: No systematic monitoring of symptoms — No systematic monitoring of symptoms will be carried out, and patients will receive the usual care. Data collection will be carried out with the assistance of a clinical research nurse up to 12 months, then under the direction of local healthcare teams at 18 months.
  Arms: Control group
Other: Systematic monitoring of symptoms — once a month, individual patient scores will be sent to dialysis staff. Any score of 3 (severe symptoms) or 4 (overwhelming) on a scale of 0 to 4, on the IPOS-Renal instrument, will be permanently reported to the referrer to trigger the patient's usual symptom management.
  Patients will complete 3 further HRQoL questionnaires at baseline, M6, M12 and M18: EQ-5D-5L, KDQoL-36, SONG Fatigue.
  A clinical research nurse will be present in half of the participating dialysis units to help patients and dialysis teams to include and follow up patients, up to 12 months. Between 12 and 18 months, data will be collected in "real life", under the guidance of local healthcare teams.
  In the other half of the dialysis units, data will be collected under the direction of the local healthcare teams, who will have to organize themselves to ensure data collection. These units will also be asked to conduct semi-structured interviews as part of the qualitative phase.
  Arms: Experimental group

SUMMARY:
In France, end-stage renal disease (ESRD) affects almost 170 people per million inhabitants every year, and 92,500 people are treated by dialysis or kidney transplantation (0.14% of the French population).

The treatment of chronic renal failure is extremely costly: 4 billion euros in 2021, i.e. 2% of health insurance expenditure, and an annual cost of 42,000 euros per patient.

The health-related quality of life (HRQoL) of dialysis patients is low, with reports of patients at 40%-60% of full health. In France, there has been a significant decrease in physical (-15.4 points) and mental (-6.9 points) component scores compared with the general population. Dialysis patients often present severe or overwhelming symptoms, which contribute to this poor HRQoL. However, in nephrology, studies have focused on survival and laboratory biomarkers, and very few interventions have been aimed at improving what was a priority for patients, i.e. treating their symptoms and improving their HRQoL. Opportunities to intervene and improve symptom management and overall HRQoL may therefore have been missed.

Ignoring patients' symptoms is an important omission. Of 28 randomized trials in primary care and oncology that measured the impact of communicating patient-reported outcomes to clinicians, 65% showed improved care processes and 47% improved health outcomes. The results of two recent randomized trials in oncology suggest that symptom monitoring can improve HRQoL and overall survival.

There is no evidence for dialysis patients, although therapeutic solutions are available in most cases.

Nephrology teams do not sufficiently recognize the prevalence, severity and negative effects of symptoms in their patients, and patients under-report their symptoms. With systematic symptom screening and automatic transmission of symptoms in the form of alerts, dialysis staff will be able to react and implement routine management to alleviate patients' symptoms.

The F-SWIFT study evaluates the hypothesis that regular symptom monitoring and feedback to hemodialysis patients and their dialysis staff improves patient HRQoL at 18 months.

In addition, the trial aims to determine whether electronic capture of patient-reported outcomes within a national dialysis patient registry is feasible and cost-effective, evaluated using consumption data from the Système National des données de Santé (SNDS) medico-administrative database.

F-SWIFT is the French part of an international project (SWIFT) initiated in Australia in 2021: Australian New Zealand Clinical Trials Registry #ACTRN12620001061921. This French part is funded by Inserm's AAP MESSIDORE 2022.

F-SWIFT is also the continuation of the pilot study n° 2021-A00776-35 accepted by the CPP EST II on 19/10/2021 and financed by the Agence de la Biomédecine (AOR 2021) in the RIPH3 category.

DETAILED DESCRIPTION:
F-SWIFT is a large-scale, multi-center, randomized controlled trial (qualitative and quantitative) nested in a national registry.

Indeed, this research project is nested in the REIN (Réseau Epidémiologique et Information en Nephrologie) registry, to which all dialysis units in France have been contributing for over 10 years. All information on the dialysis units and the patients included is taken directly from the register. The field presence of REIN's clinical research officers ensures the quality of the data routinely collected for the registry, and reused in this project.

The F-SWIFT project includes a process analysis to support the transferability of F-SWIFT in the event of proven effectiveness, with a view to large-scale deployment.

Data analysis will be carried out by a biostatistician and Human and Social Sciences engineers from CIC 1433 Epidémiologie Clinique at CHRU Nancy.

In accordance with the third paragraph of article 56 of the French Data Protection Act, the presentation of the results of data processing may under no circumstances allow direct or indirect identification of the persons involved in the research.

Experimental group

* Quarterly measurement for 18 months of patients' symptoms using the IPOS-Renal questionnaire, which will be systematically reported to professionals.
* Measurement every 6 months for 18 months of patients' health-related HRQoL using the EQ-5D-5L (European Quality of Life 5 Dimensions 5 Level Version), KDQoL-36 (Kidney Disease and Quality of Life™ Short Form) and SONG-Fatigue (Stadardised Outcomes in NephroloGy Fatigue) questionnaires.

Control group

* No systematic symptom monitoring will be organized, and patients will receive usual care.
* Measurement every 6 months for 18 months of health-related HRQoL using the EQ-5D-5L, KDQoL-36 and SONG-Fatigue questionnaires.

Process evaluation phase

Quantitative component

For all dialysis units included in the experimental arm:

The REIN registry will provide data on: legal status, volume of patients managed, treatment options offered. The REIN registry will also provide data on patients in these units: age, sex, comorbidity, length of time on dialysis and dialysis treatment modality.

For patients at inclusion, an ad hoc questionnaire will be added on electronic equipment at home, which includes the availability and use of a laptop, desktop, tablet, cell phone and broadband internet subscription.

Per unit, every 3 months, loyalty criteria (% of patients having completed the IPOS-Renal questionnaire) and dose criteria (cumulative number of completed IPOS-Renal questionnaires) will be collected.

Based on the reimbursement list provided by the health insurance (data extracted from the REIN register linked to the SNDS), changes in prescribing practices will be studied (prescription of drugs and supportive care, in particular dietary, psychological and sports care). The before-and-after trends will be analyzed one year after the end of the study in the unit (remote evaluation), since the data are only consolidated at that time.

Qualitative component:

Three months after the start of the study, from among the units in the experimental group meeting the condition without external assistance from the Clinical Research Nurse (CRN) to collect data, five units will be selected following an extreme case sampling (2 with the highest level, 1 with a standard level and 2 with the lowest level of intervention application) to conduct semi-structured interviews.

At this stage, the research team will focus on organizational and implementation factors to provide information for the scientific committee, which will be responsible for decisions to adapt the F-SWIFT intervention and improve its effectiveness. After three months of fine-tuning the intervention, the research team will carry out a second wave of qualitative process evaluation to (re)test the intervention in five other units.

Semi-structured individual interviews will therefore be conducted with patients and healthcare professionals (nurses and doctors) on the basis of a guide developed to gather perceptual data on how contextual characteristics affect the effective implementation and outcomes of the F-SWIFT intervention.

Participants in the individual semi-structured interview will receive an e-mail from an engineer in the humanities and social sciences, informing them of the date and time of the appointment, as well as the connection link if the interview takes place remotely.

ELIGIBILITY:
Inclusion Criteria:

Symptom collection phase

The inclusion criteria for patients are as follows:

* Individuals who have received full information on the organization of the research and who have not objected to their participation and to the use of their data.
* Adults aged 18 and over
* Patients with end-stage renal disease treated by dialysis in participating dialysis units
* Patients able to answer questionnaires

Process evaluation phase

The inclusion criteria for healthcare professionals are as follows:

* Individuals who have received full information on the organization of the research and who have not objected to their participation and to the use of their data.
* Patients with end-stage renal disease treated by dialysis in participating dialysis units.
* Doctors and nurses working in the dialysis unit taking part in the study.

Exclusion Criteria:

The non-inclusion criteria for patients are as follows:

* Minors
* Patients under legal protection, guardianship or curatorship
* Patient not communicating or unable to give consent
* Patient not being treated in a dialysis unit participating in the study
* Patients being treated temporarily in a participating dialysis unit (respite care, vacationers, etc.)
* Patient with cognitive disorders
* Patient unable or unwilling to answer questionnaires

The non-inclusion criteria for healthcare professionals are as follows:

* Non-voluntary healthcare professional
* Healthcare professional not working in the participating facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2293 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life over 12 months, measured by the physical health score of the validated Kidney Disease and Quality of Life™ Short Form (KDQoL-36) questionnaire. | 12 months
  KDQoL-36 Short form assesses quality of life over the past 4 weeks. Physical health score ranges from 0=Worst quality of life to 100=Best quality of life

SECONDARY OUTCOMES:
Respondents' perceptions of the impact of the system's implementation and changes in practices | 3 months
  semi-structured interviews analyzed by NVivo
12-month survival measured using REIN registry data | 12 months
  percentage (0 to 100%) of patients alive at 12 months
Questionnaire completion rates for different arms and periods. | 12 months
  Percentage (0 to 100%) of questionnaire completed
Severity of symptoms measured using the IPOS Renal (Integrated Palliative Outcome Score Renal) questionnaires | 18 months
  Describe the severity of symptoms and their relationship to comorbidities in dialysis patients in the intervention group.
Severity of symptoms measured using the SONG fatigue (Stadardised Outcomes in NephroloGy Fatigue) questionnaires | 18 months
  Describe the severity of symptoms and their relationship to comorbidities in dialysis patients in the intervention group.
  Song Fatigue : Minimum value: not at all maximum value: extremely Maximum value means a worse result
Severity of symptoms measured using the SONG fatigue (Stadardised Outcomes in NephroloGy Fatigue) questionnaires | 18 months
  Evaluate the effectiveness of the intervention on the mental health score of the validated KDQoL-36 questionnaire.
  Song Fatigue : Minimum value: not at all maximum value: extremely Maximum value means a worse result
12-month survival measured using REIN data | 18 months
  Evaluate the effectiveness of the intervention at 18 months and the sustainability of practices based on the indicators used in the main objective and secondary objectives 2, 3 and 6.
Numbers of care consumption, including hospitalizations, drugs, prescriptions for biological and imaging tests, based on SNDS data. | 18 months
  Evaluate the effectiveness of the intervention at 18 months and the sustainability of practices based on the indicators used in the main objective and secondary objectives 2, 3 and 6.
Incremental cost between intervention and no-intervention groups related to the quality-adjusted life-year differential assessed by the evolution of utility at 12 months measured by the EQD5D-5L questionnaire. | 18 months
  Evaluate the effectiveness of the intervention at 18 months and the sustainability of practices based on the indicators used in the main objective and secondary objectives 2, 3 and 6.
Duration of dialysis measured using REIN registry data. | 18 months
  Evaluate the effectiveness of the intervention at 18 months and the sustainability of practices based on the indicators used in the main objective and secondary objectives 2, 3 and 6.
Frequency of dialysis measured using REIN registry data. | 18 months
  Evaluate the effectiveness of the intervention at 18 months and the sustainability of practices based on the indicators used in the main objective and secondary objectives 2, 3 and 6.
Number of dialysis stops measured using REIN registry data. | 18 months
  Evaluate the effectiveness of the intervention at 18 months and the sustainability of practices based on the indicators used in the main objective and secondary objectives 2, 3 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Francis GUILLEMIN, MD, PhD, Principal Investigator — Centre d'Investigation Clinique - Epidémiologie Clinique 1433
Locations (1):
- Ostermann, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wyld M, Morton RL, Hayen A, Howard K, Webster AC. A systematic review and meta-analysis of utility-based quality of life in chronic kidney disease treatments. PLoS Med. 2012;9(9):e1001307. doi: 10.1371/journal.pmed.1001307. Epub 2012 Sep 11. PMID 22984353
- [Background] Janssen DJ, Spruit MA, Wouters EF, Schols JM. Daily symptom burden in end-stage chronic organ failure: a systematic review. Palliat Med. 2008 Dec;22(8):938-48. doi: 10.1177/0269216308096906. Epub 2008 Sep 18. PMID 18801874
- [Background] Tong A, Chando S, Crowe S, Manns B, Winkelmayer WC, Hemmelgarn B, Craig JC. Research priority setting in kidney disease: a systematic review. Am J Kidney Dis. 2015 May;65(5):674-83. doi: 10.1053/j.ajkd.2014.11.011. Epub 2015 Jan 10. PMID 25582284
- [Background] You AS, Kalantar SS, Norris KC, Peralta RA, Narasaki Y, Fischman R, Fischman M, Semerjian A, Nakata T, Azadbadi Z, Nguyen DV, Kalantar-Zadeh K, Rhee CM. Dialysis symptom index burden and symptom clusters in a prospective cohort of dialysis patients. J Nephrol. 2022 Jun;35(5):1427-1436. doi: 10.1007/s40620-022-01313-0. Epub 2022 Apr 16. PMID 35429297
- [Background] Fletcher BR, Damery S, Aiyegbusi OL, Anderson N, Calvert M, Cockwell P, Ferguson J, Horton M, Paap MCS, Sidey-Gibbons C, Slade A, Turner N, Kyte D. Symptom burden and health-related quality of life in chronic kidney disease: A global systematic review and meta-analysis. PLoS Med. 2022 Apr 6;19(4):e1003954. doi: 10.1371/journal.pmed.1003954. eCollection 2022 Apr. PMID 35385471
- [Background] Kalantar-Zadeh K, Lockwood MB, Rhee CM, Tantisattamo E, Andreoli S, Balducci A, Laffin P, Harris T, Knight R, Kumaraswami L, Liakopoulos V, Lui SF, Kumar S, Ng M, Saadi G, Ulasi I, Tong A, Li PK. Patient-centred approaches for the management of unpleasant symptoms in kidney disease. Nat Rev Nephrol. 2022 Mar;18(3):185-198. doi: 10.1038/s41581-021-00518-z. Epub 2022 Jan 3. PMID 34980890
- [Background] Raghavan D, Holley JL. Conservative Care of the Elderly CKD Patient: A Practical Guide. Adv Chronic Kidney Dis. 2016 Jan;23(1):51-6. doi: 10.1053/j.ackd.2015.08.003. PMID 26709063
- [Background] Davison SN, Levin A, Moss AH, Jha V, Brown EA, Brennan F, Murtagh FE, Naicker S, Germain MJ, O'Donoghue DJ, Morton RL, Obrador GT; Kidney Disease: Improving Global Outcomes. Executive summary of the KDIGO Controversies Conference on Supportive Care in Chronic Kidney Disease: developing a roadmap to improving quality care. Kidney Int. 2015 Sep;88(3):447-59. doi: 10.1038/ki.2015.110. Epub 2015 Apr 29. PMID 25923985
- [Background] Greenham L, Bennett PN, Dansie K, Viecelli AK, Jesudason S, Mister R, Smyth B, Westall P, Herzog S, Brown C, Handke W, Palmer SC, Caskey FJ, Couchoud C, Simes J, McDonald SP, Morton RL. The Symptom Monitoring with Feedback Trial (SWIFT): protocol for a registry-based cluster randomised controlled trial in haemodialysis. Trials. 2022 May 19;23(1):419. doi: 10.1186/s13063-022-06355-0. PMID 35590395
- [Background] Viecelli AK, Duncanson E, Bennett PN, D'Antoine M, Dansie K, Handke W, Tong A, Palmer S, Jesudason S, McDonald S, Morton RL; Symptom Monitoring With Feedback Trial (SWIFT) Investigators. Perspectives of Patients, Nurses, and Nephrologists About Electronic Symptom Monitoring With Feedback in Hemodialysis Care. Am J Kidney Dis. 2022 Aug;80(2):215-226.e1. doi: 10.1053/j.ajkd.2021.12.007. Epub 2022 Jan 25. PMID 35085687
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Lockwood MB, Lash JP, Pauls H, Chung SY, Samra M, Ryan C, Park C, DeVon H, Bronas UG. Physical Symptom Cluster Subgroups in Chronic Kidney Disease. Nurs Res. 2020 Mar/Apr;69(2):100-108. doi: 10.1097/NNR.0000000000000408. PMID 31714343
- [Background] Abdel-Kader K, Unruh ML, Weisbord SD. Symptom burden, depression, and quality of life in chronic and end-stage kidney disease. Clin J Am Soc Nephrol. 2009 Jun;4(6):1057-64. doi: 10.2215/CJN.00430109. Epub 2009 May 7. PMID 19423570
- [Background] Kalantar-Zadeh K, Li PK, Tantisattamo E, Kumaraswami L, Liakopoulos V, Lui SF, Ulasi I, Andreoli S, Balducci A, Dupuis S, Harris T, Hradsky A, Knight R, Kumar S, Ng M, Poidevin A, Saadi G, Tong A; World Kidney Day Steering Committee. Living well with kidney disease by patient and care-partner empowerment: Kidney health for everyone everywhere. Saudi J Kidney Dis Transpl. 2021 Mar-Apr;32(2):289-297. doi: 10.4103/1319-2442.335439. PMID 35017321
- [Background] Jais JP, Lobbedez T, Couchoud C. [Survival of patients with End Stage Kidney Disease]. Nephrol Ther. 2023 Aug 28;18(S2):35-39. doi: 10.1016/S1769-7255(22)00565-X. French. PMID 37638506
- [Background] Vaismoradi M, Turunen H, Bondas T. Content analysis and thematic analysis: Implications for conducting a qualitative descriptive study. Nurs Health Sci. 2013 Sep;15(3):398-405. doi: 10.1111/nhs.12048. Epub 2013 Mar 11. PMID 23480423